CLINICAL TRIAL: NCT03794713
Title: A Randomized, Two-arm, Open Label Study to evalUate the Effect of a Smart Phone-based Patient Support Tool On Patient AdheRence of Treatment in Stable Angina Patients Prescribed Beta-blockers in China (SUPPORT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Dr, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPPORT V1.0
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Adrenergic Beta-Antagonists; Stable Angina Pectoris; Medication Adherence; Mobile Applications
Keywords: beta-blocker; Stable Angina Pectoris; Patient support tool; Adherence
MeSH Terms: conditions — Angina, Stable; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient support tool group (Experimental): Subjects were managed the HR by using the Patient Support Tool through a smart phone application and a wristband and be guided by physicians
  Interventions: Device: Patient support tool
- Control group (No Intervention): Subjects were received a usual patient care at baseline, which left to the discretion of physicians, without any specific intervention at follow-up period

INTERVENTIONS:
Device: Patient support tool — The patient support tool, a software app installed on the smart phones plus a wrist connected to the smart phones by Bluetooth. The wrist could monitor the pulse, which was recorded to the app in the smart phone. Meanwhile, the app could inform to patients about the importance of medication, remind on the medicine intake, share the patients' data with themselves, and warn the patients if the wrist don't wear.
  Arms: Patient support tool group

SUMMARY:
The present study aims to enhance the adherence of beta-blockers by Patient Support Tool through a smart phone application and a wristband, subsequently reduce the risk of angina attacks in patients with stable angina pectoris.

DETAILED DESCRIPTION:
To control heart rate in terms of guidelines in patients with stable angina pectoris reduces risk of cardiovascular events, rehospitalization, and death effectively. Using beta blockers is an efficient therapy to management the HR in SAP patients. However, the recent epidemiological studies have provided evidences that the rate of beta blocker prescribed and used was inadequate, as the first-line therapy to CAD patients with the usage rate less than 30%. Several studies showed that with a reminder supported by smart phones and wearable devices, the adherence of management of patients with chronic disease could be improved significantly.Thus,the present study aims to enhance the adherence of beta-blockers by Patient Support Tool through a smart phone application and a wristband, subsequently reduce the risk of angina attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Stable angina pectoris;
3. Indicated for beta blockers;
4. HR ≥ 60bpm;
5. Patient must have a smart phone that is compatible with the Patient support tool at their disposal and are comfortable with using of interactive smart phone applications. The required specification for the phone will be determined after completed testing;
6. Ability to read, understand and write Chinese;
7. Beta-blockers naïve or with no Beta-blocker use during the last 1 month.

Exclusion Criteria:

1. Previous myocardial infarction during the recent 1 year;
2. Cardiac shock or unstable heart failure (NYHA III);
3. SBP<100 mmHg;
4. Sick sinus syndrome;
5. II-III degree atrioventricular block;
6. Existing contraindication for Beta-blockers or allergic to beta-blockers;
7. Participation in another clinical study with a beta blocker during the last 3 months;
8. Inability to sign the informed consent form;
9. Females during pregnancy and lactation and women of child bearing potential planning to be pregnant within 24 weeks.;
10. Patients who withdraw from this study for any reason cannot re-enter the study;
11. Life expectancy < 1 year;
12. Severe asthma or COPD;
13. Severe peripheral vascular disease;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to beta-blockers | 24 weeks
  To evaluate the effect of Patient Support Tool through a smart phone application and a wristband on adherence to beta-blockers in patients with stable coronary artery disease.Duration of treatment-defined as the days the Patient has taken beta-blockers followed the advice of doctors during the 24-week follow up.

SECONDARY OUTCOMES:
Impact of resting heart rate | 24 weeks
  To evaluate the impact of the Patient Support Tool on rHR (resting heart rate).The difference of the average rHR change from baseline between 2 groups.
Impact of angina attacks | 24 weeks
  To evaluate the impact of the Patient Support Tool on Angina attacks. The difference of the score change of Seattle angina Questionnaire.
Major adverse cardiovascular events | 24 weeks
  To evaluate the impact of the Patient Support Tool on major adverse cardiovascular events (MACE), a composite of cardiac death, myocardial infarction, stroke, and revascularization.

IPD SHARING:
Plan to Share IPD: No